CLINICAL TRIAL: NCT00544830
Title: Androgen Deprivation and Localized Radiotherapy to Metastases in Patients With Oligometastatic Hormone - Sensitive Prostate Cancer
Brief Title: Hormone Therapy and Intensity-Modulated Radiation Therapy in Treating Patients With Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05190; NCI-2010-00425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 05190 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2022-04-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: PSA Level Greater Than Two; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — bicalutamide; Goserelin; Radiotherapy, Intensity-Modulated; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (androgen therapy, radiation therapy) (Experimental): ADT: Patients not currently on ADT receive goserelin acetate SC or leuprolide acetate via injection once every 4 or 12 weeks and bicalutamide PO QD. Treatment repeats every 12 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients already receiving ADT at the time of enrollment continue treatment until they have received 36 weeks of therapy.
  RADIATION THERAPY: Patients achieving PSA normalization after initiation of androgen deprivation therapy undergo intensity-modulated radiation therapy daily for 2-7 weeks during or after completion of androgen deprivation therapy.
  Interventions: Drug: Bicalutamide; Drug: Goserelin Acetate; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leuprolide Acetate — Given via injection
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur

SUMMARY:
This phase II trial studies how well hormone therapy and intensity-modulated radiation therapy work in treating patients with prostate cancer that has spread to other places in the body. Androgens can cause the growth of prostate cancer cells. Anti-hormone therapy using goserelin, leuprolide acetate, or bicalutamide, may lessen the amount of androgens made by the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving hormone therapy and intensity-modulated radiation therapy may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the time to prostate-specific antigen (PSA) relapse in patients with oligometastatic (=< 5 lesions) hormone-sensitive prostate cancer treated with 36 weeks of androgen deprivation therapy and localized radiotherapy to all known tumor sites.

II. To assess the prostate-specific-antigen (PSA) and objective response rate to treatment with 36 weeks of androgen deprivation and localized radiotherapy in patients with oligometastatic hormone-sensitive prostate cancer.

III. To assess the toxicity of 36 weeks of androgen deprivation and localized radiation therapy to oligometastases in patients with oligometastatic hormone-sensitive prostate cancer.

IV. In appropriate situations evaluate the feasibility and toxicities of using helical tomotherapy image-guided intensity-modulated radiation therapy (IMRT) to treat oligometastatic sites.

OUTLINE:

ANDROGEN DEPRIVATION THERAPY (ADT): Patients not currently on ADT receive goserelin acetate subcutaneously (SC) or leuprolide acetate via injection once every 4 or 12 weeks and bicalutamide orally (PO) once daily (QD). Treatment repeats every 12 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients already receiving ADT at the time of enrollment continue treatment until they have received 36 weeks of therapy.

RADIATION THERAPY: Patients achieving PSA normalization after initiation of androgen deprivation therapy undergo intensity-modulated radiation therapy daily for 2-7 weeks during or after completion of androgen deprivation therapy.

After completion of study treatment, patients are followed up every 4 weeks for 2 years, then every 3 months after year 2, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven diagnosis of adenocarcinoma of the prostate stage N1, N2, N3, M1a, M1b, M1c with =< 5 metastatic lesions; if the diagnosis of metastasis in the lymph node is based solely on imaging computed tomography (CT) scan or magnetic resonance imaging (MRI), the longitudinal diameter of the lymph node has to be >= 2.0 cm; if the lymph node is positive on positron emission tomography (PET) or ProstaScint scan, the longitudinal diameter of the lymph node on CT scan or MRI has to be >= 1.5 cm
* Patients who have measurable disease must have had X-rays, scans or physical examination used for tumor measurement completed within 28 days prior to registration; patients must have non-measurable disease assessed within 42 days prior to registration
* Patients must have had documented PSA of > 2 prior to onset of androgen deprivation
* Patients might have received up to 36 weeks of adjuvant androgen deprivation therapy and up to 36 weeks of androgen deprivation therapy for metastatic disease prior to enrollment to this study; patients may be on androgen deprivation for metastatic disease at the time of enrollment to the protocol; adjuvant therapy must have been completed at least 2 years before androgen deprivation for metastatic disease and patients must remain hormone sensitive
* Prior radiation therapy for metastatic disease is not allowed
* Prior chemotherapy for metastatic disease is not allowed; prior neoadjuvant and adjuvant chemotherapy is allowed; patients must have recovered from all acute side-effects related to previous systemic therapy
* Patients are allowed to receive one prior systemic non-chemotherapeutic treatment (i. e. immunotherapy, receptor tyrosine kinase inhibitor, antiangiogenic agent, differentiation agent) for recurrent or metastatic disease; patients must have recovered from all acute side-effects related to previous systemic therapy
* Use of bisphosphonates is allowed at the discretion of treating physician
* Patients must be capable of understanding the nature of the trial and must give written informed consent
* Patients must have a World Health Organization (WHO) performance status of 0, 1, or 2

Exclusion Criteria:

* Patients with unstable or severe intercurrent medical conditions or active, uncontrolled infection
* Patients with a history of orchiectomy
* Patients undergoing therapy with other investigational agents; patients must have recovered from all acute effects of previously administered investigational agents and sufficient time must have elapsed since last administration to ensure the drug interactions not occur during this study
* Patients with a history of brain metastases or who currently have treated or untreated brain metastases
* Patients who have demonstrated refractoriness to hormone therapy with luteinizing hormone-releasing hormone (LHRH) agonist; refractoriness is defined as occurrence of one of the following while on therapy with LHRH agonist: increase in PSA by 25% over baseline (to at least > 2 ng/ml) on two consecutive PSA measurements, 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, clear worsening of any non-measurable disease, reappearance of any lesion that had disappeared, appearance of any new lesion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-07-18 (Actual); Primary Completion 2011-03-16 (Actual); Study Completion 2026-03-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cy A Stein, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was consented on July 18, 2006. The last eligible patient was consented on August 25, 2010. Patients were recruited at City of Hope National Medical Center.
Groups:
- Treatment (Androgen Therapy, Radiation Therapy): ADT: Patients not currently on ADT receive goserelin acetate SC or leuprolide acetate via injection once every 4 or 12 weeks and bicalutamide PO QD. Treatment repeats every 12 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients already receiving ADT at the time of enrollment continue treatment until they have received 36 weeks of therapy.
  RADIATION THERAPY: Patients achieving PSA normalization after initiation of androgen deprivation therapy undergo intensity-modulated radiation therapy daily for 2-7 weeks during or after completion of androgen deprivation therapy.
  Bicalutamide: Given PO
  Goserelin Acetate: Given SC
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Leuprolide Acetate: Given via injection
Period: Overall Study
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 66.9 [49.5 to 79.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants] — City of Hope National Medical Center, Duarte, CA USA
  Participants
    United States | 29
Baseline Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/ml] — The number of patients reaching a nadir of PSA < 0.2 will be reported in the results.
  ng/ml | 11.4 [1 to 74.5]
Metastases limited to pelvic lymph nodes [Count of Participants; unit: Participants] — Count of patients with metastases limited to pelvic lymph nodes. This baseline is referenced in the results section.
  Participants | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate-specific Antigen (PSA) Relapse
Description: Time from the date of the last dose of bicalutamide or the last day of radiation therapy (whichever comes later) until the date criteria are met for PSA relapse. PSA relapse after completion of initial 36 weeks of androgen deprivation therapy is defined as an increase in PSA value to above pre-therapy level, or to > 10, whichever is smaller. For example, a patient with pre-treatment PSA level of 40 will resume androgen deprivation therapy when PSA level is > 10, while a patient with pre-treatment PSA level of 3 will resume androgen deprivation therapy when PSA level is > 3.
Time Frame: End-of-therapy until PSA reached pre-treatment level or 10 (whichever was lower)
Population: Metastatic prostate cancer patients treated with androgen deprivation.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 29
month | 16.5 [14.0 to 34.3]

2. Secondary Outcome: Patients Who Achieved PSA Nadir of < 0.2 at 36 Weeks.
Description: Number of Patients who achieved PSA nadir of < 0.2 at 36 weeks.
Time Frame: During the time period between on-study PSA to off-study PSA, up to 36 weeks.
Population: Patients who achieved PSA nadir of < 0.2 at 36 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 29
Participants | 25

3. Secondary Outcome: Rate of Treatment Failure (no PSA Threshold Below 4 ng/dl, or no PSA Below Baseline Level Before LHRH Treatment).
Description: Treatment failures: Count and percent of patients NOT reaching PSA concentration in serum either below 4 ng/dl or below baseline before LHRH treatment .
Time Frame: Off-treatment PSA measurement date minus on-study PSA measurement date, up to 36 weeks.
Population: Metastatic prostate cancer patients treated with androgen deprivation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 29
Participants | 15

4. Secondary Outcome: Length of Follow-up
Description: Length of follow-up in weeks to off-study date. Patients are treated for 36 weeks (+/- 2 weeks) with androgen deprivation therapy. Patients are evaluated for disease on day 1 of each of three 12-week cycles. After the last cycle of anti-androgen therapy, patients are assessed every four weeks until PSA relapse occurs, up to 264.8 weeks (61.4 months; 5.1 years). Patients will remain off-treatment until they meet the criteria for re-treatment with androgen deprivation therapy, whereupon they will be taken off of the protocol. After patients are taken off protocol, we will do a chart review for long-term outcomes.
Time Frame: Patients are evaluated for disease on day 1 of each of three 12-week cycles. After the last cycle of anti-androgen therapy, patients are assessed every four weeks until PSA relapse occurs, up to 61.4 months
Population: Patients with hormone sensitive prostate cancer
Measure: Median (Full Range); unit: week
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 29
week | 111.4 [58.1 to 264.8]

5. Secondary Outcome: Count of Patients Remaining Off of Therapy
Description: Patients who remained off of therapy, in remission, out of the number of patients with metastases limited to pelvic lymph nodes.
Time Frame: after 36 week LHRH treatment window.
Population: Patients with metastases limited to pelvic lymph nodes
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 8
Participants | 7

6. Secondary Outcome: Follow-up of the 8 Patients With Metastases Limited to Pelvic Lymph Nodes.
Description: Length of follow-up of the 8 patients with metastases limited to pelvic lymph nodes, months. Patients are followed on day one of each of three 12-week periods. After completion of therapy, patients are followed every four weeks until PSA relapse, up to 46.4 months.
Time Frame: Patients are followed on day one of each of three 12-week periods. After completion of therapy, patients are followed every four weeks until PSA relapse, up to 46.4 months.
Population: Patients with metastases limited to pelvic lymph nodes.
Measure: Median (Full Range); unit: month
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 8
month | 14.7 [9.2 to 46.4]

7. Secondary Outcome: CR Without ADT in Patients With Metastases Limited to Pelvic Lymph Nodes.
Description: Number of patients remaining in complete remission without androgen deprivation therapy in patients with metastases limited to pelvic lymph nodes.
Time Frame: after 36 weeks of LHRH therapy.
Population: Patients with metastases limited to pelvic lymph nodes.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Number analyzed (Participants) | 8
Participants | 4

ADVERSE EVENTS:
Arm/Group | Treatment (Androgen Therapy, Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Androgen Therapy, Radiation Therapy) (N=29)
10012727 -- Diarrhea (Gastrointestinal disorders) | 1 (1)
10010300 -- Confusion (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Androgen Therapy, Radiation Therapy) (N=29)
10019483 -- Hemoglobin decreased (Blood and lymphatic system disorders) | 20 (20)
10019483 -- Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
10003658 -- Atrial fibrillation (Cardiac disorders) | 1 (1)
10003668 -- Atrial tachycardia (Cardiac disorders) | 1 (1)
10040741 -- Sinus bradycardia (Cardiac disorders) | 6 (6)
10019246 -- Hearing loss (Ear and labyrinth disorders) | 1 (1)
10014695 -- Endocrine disorder (Endocrine disorders) | 1 (1)
10000081 -- Abdominal pain (Gastrointestinal disorders) | 1 (1)
10010774 -- Constipation (Gastrointestinal disorders) | 3 (3)
10012727 -- Diarrhea (Gastrointestinal disorders) | 15 (15)
10013950 -- Dysphagia (Gastrointestinal disorders) | 2 (2)
10015461 -- Esophagitis (Gastrointestinal disorders) | 1 (1)
10016766 -- Flatulence (Gastrointestinal disorders) | 3 (3)
10017944 -- Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4)
10018286 -- Gingival pain (Gastrointestinal disorders) | 1 (1)
10019611 -- Hemorrhoids (Gastrointestinal disorders) | 8 (8)
10028813 -- Nausea (Gastrointestinal disorders) | 4 (4)
10036774 -- Proctitis (Gastrointestinal disorders) | 1 (1)
10036787 -- Proctoscopy abnormal (Gastrointestinal disorders) | 1 (1)
10038064 -- Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
10038072 -- Rectal pain (Gastrointestinal disorders) | 1 (1)
10047700 -- Vomiting (Gastrointestinal disorders) | 2 (2)
10056848 -- Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
10065709 -- Rectal necrosis (Gastrointestinal disorders) | 1 (1)
10012727 -- Diarrhea (Gastrointestinal disorders) | 2 (2)
10028813 -- Nausea (Gastrointestinal disorders) | 1 (1)
10008479 -- Chest pain (General disorders) | 2 (2)
10016256 -- Fatigue (General disorders) | 14 (14)
10016558 -- Fever (General disorders) | 1 (1)
10033371 -- Pain (General disorders) | 1 (1)
10050068 -- Edema limbs (General disorders) | 4 (4)
90004082 -- Pain (General disorders) | 3 (3)
10008531 -- Chills (General disorders) | 1 (1)
10016558 -- Fever (General disorders) | 1 (1)
90004082 -- Pain (General disorders) | 1 (1)
10020751 -- Hypersensitivity (Immune system disorders) | 1 (1)
10021789 -- Infection (Infections and infestations) | 1 (1)
90031098 -- Upper respiratory infection (Infections and infestations) | 1 (1)
90031102 -- Urinary tract infection (Infections and infestations) | 1 (1)
10061103 -- Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
10065892 -- Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
10061103 -- Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
10001551 -- Alanine aminotransferase increased (Investigations) | 6 (6)
10001675 -- Alkaline phosphatase increased (Investigations) | 1 (1)
10003481 -- Aspartate aminotransferase increased (Investigations) | 9 (9)
10011349 -- Creatine phosphokinase increased (Investigations) | 2 (2)
10011368 -- Creatinine increased (Investigations) | 2 (2)
10025256 -- Lymphocyte count decreased (Investigations) | 18 (18)
10029366 -- Neutrophil count decreased (Investigations) | 2 (2)
10035528 -- Platelet count decreased (Investigations) | 12 (12)
10040190 -- Serum cholesterol increased (Investigations) | 2 (2)
10047896 -- Weight gain (Investigations) | 2 (2)
10048552 -- Leukocyte count decreased (Investigations) | 18 (18)
10024384 -- Leukopenia (Investigations) | 2 (2)
10025327 -- Lymphopenia (Investigations) | 1 (1)
10035528 -- Platelet count decreased (Investigations) | 1 (1)
10002646 -- Anorexia (Metabolism and nutrition disorders) | 2 (2)
10005557 -- Blood glucose increased (Metabolism and nutrition disorders) | 10 (10)
10012174 -- Dehydration (Metabolism and nutrition disorders) | 1 (1)
10040123 -- Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
10040175 -- Serum calcium increased (Metabolism and nutrition disorders) | 6 (6)
10040268 -- Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2)
10040336 -- Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
10040378 -- Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
10040379 -- Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
10040405 -- Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
10040424 -- Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (2)
10054863 -- Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
10021018 -- Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
10003246 -- Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
10003988 -- Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
10006002 -- Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10023222 -- Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
10028411 -- Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
10028836 -- Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
10031282 -- Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3)
10033425 -- Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
10013573 -- Dizziness (Nervous system disorders) | 2 (2)
10019211 -- Headache (Nervous system disorders) | 2 (2)
10029298 -- Neurological disorder NOS (Nervous system disorders) | 1 (1)
10034620 -- Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
10002855 -- Anxiety (Psychiatric disorders) | 4 (4)
10012378 -- Depression (Psychiatric disorders) | 1 (1)
10022437 -- Insomnia (Psychiatric disorders) | 2 (2)
10024419 -- Libido decreased (Psychiatric disorders) | 2 (2)
10011781 -- Cystitis (Renal and urinary disorders) | 1 (1)
10019591 -- Hemorrhage urinary tract (Renal and urinary disorders) | 4 (4)
10037020 -- Protein urine positive (Renal and urinary disorders) | 2 (2)
10038435 -- Renal failure (Renal and urinary disorders) | 1 (1)
10046461 -- Urethral pain (Renal and urinary disorders) | 4 (4)
10046539 -- Urinary frequency (Renal and urinary disorders) | 22 (22)
10046543 -- Urinary incontinence (Renal and urinary disorders) | 6 (6)
10046555 -- Urinary retention (Renal and urinary disorders) | 4 (4)
10046694 -- Urogenital disorder (Renal and urinary disorders) | 2 (2)
10046694 -- Urogenital disorder (Renal and urinary disorders) | 1 (1)
10034310 -- Penile pain (Reproductive system and breast disorders) | 1 (1)
10036968 -- Prostatic pain (Reproductive system and breast disorders) | 1 (1)
10061461 -- Erectile dysfunction (Reproductive system and breast disorders) | 10 (10)
10018801 -- Gynecomastia (Reproductive system and breast disorders) | 1 (1)
10011224 -- Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10013963 -- Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10034844 -- Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10035598 -- Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10047681 -- Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10001760 -- Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
10013786 -- Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
10037087 -- Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
10037853 -- Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (5)
10040831 -- Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
10040865 -- Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
10020407 -- Hot flashes (Vascular disorders) | 18 (18)
10020772 -- Hypertension (Vascular disorders) | 1 (1)
10021097 -- Hypotension (Vascular disorders) | 1 (1)
10020407 -- Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT00544830/Prot_SAP_000.pdf